CLINICAL TRIAL: NCT03971032
Title: A Development of an In-vitro Real-time System Based on Tissue Smears to Identify Malignancy During Hysteroscopic Procedure Using FTIR-ATR Spectroscopy
Brief Title: An In-vitro Real-time System Based on Tissue Smears to Identify Malignancy During Hysteroscopic Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0098-18
Record Dates: First submitted 2019-05-01; First posted 2019-06-03 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Uterine Cervical Neoplasm; Uterine Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women undergoing hysteroscopy (Other): Women presenting with abnormal bleeding, abnormal cervical or uterine findings who have consented to undergo hysteroscopy
  Interventions: Procedure: Hysteroscopy; Device: Infrared Spectroscopy

INTERVENTIONS:
Procedure: Hysteroscopy — Diagnostic procedure
Device: Infrared Spectroscopy — This device uses spectral absorption of the tissue taken during hysteroscopy to determine immediate diagnosis of malignancy

SUMMARY:
The aim of the current study is to develop a near real-time system using infrared spectroscopy, that will evaluate the histological specimen that was removed from the uterine cavity during the hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hysteroscopy

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2019-12-31 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of infrared spectroscopy with routine histopathology | 3 years
  Tissue smears that have undergone infrared spectroscopy during hysteroscopy will have a different spectral absorption than healthy tissue, thus indicating malignancy. These results will be compared to the results of routine histopathology to determine accuracy of spectroscopy to indicate malignancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No